CLINICAL TRIAL: NCT05277675
Title: A Prospective Study of Radiofrequency Ablation Combined With Systematic Neoadjuvant Therapy in the Treatment of Recurrent Hepatocellular Carcinoma
Brief Title: Radiofrequency Ablation Plus Systematic Neoadjuvant Therapy for Recurrent Hepatocellular Carcinoma (RANT Study)
Acronym: RANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, fengkai, Associate Professor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (A)KY2021083
Record Dates: First submitted 2022-02-27; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma Recurrent
Keywords: immune checkpoint inhibitors; targeted therapy; neoadjuvant therapy; radiofrequency ablation; hepatocellular carcinoma; recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — tislelizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant therapy+ RFA (Experimental): After confirmation of HCC recurrence by imaging exam, subjects will receive neoadjuvant therapy (immune checkpoint inhibitors + targeted therapy) and then RFA
  Interventions: Drug: Tislelizumab/Sintilimab+Lenvatinib/Bevacizumab; Procedure: RFA
- RFA alone (Active Comparator): After confirmation of HCC recurrence by imaging exam, subjects will receive RFA treatment only.
  Interventions: Procedure: RFA

INTERVENTIONS:
Drug: Tislelizumab/Sintilimab+Lenvatinib/Bevacizumab — Immune checkpoint inhibitor (tislelizumab/sintilimab) combined with anti-angiogenic drugs (lenvatinib/bevacizumab) used as neoadjuvant therapy
  Arms: Neoadjuvant therapy+ RFA
Procedure: RFA — RFA will be performed in a percutaneous way guided contrast enhanced ultrasound.

SUMMARY:
1. To compare systemic neoadjuvant therapy (combination of immune checkpoint inhibitors and anti-angiogenic drugs (short for "targeted-immune therapy") combined with radiofrequency ablation (RFA) and RFA alone in the treatment of recurrent hepatocellular carcinoma(HCC) in 1-year recurrence-free survival (RFS) and overall survival (OS)
2. To evaluate the clinical value of systemic neoadjuvant therapy (i.e. immune checkpoint inhibitors and targeted therapy) combined with RFA in the treatment of recurrent HCC, as well as the safety and efficacy of this strategy.

DETAILED DESCRIPTION:
RFA is an important minimally invasive approach for recurrent HCC treatment, but is hampered by the high recurrence rate and limited ablation volume for the tumor. Therefore, the key to improving the efficacy of RFA is to maximize the complete ablation zone of tumor lesions and the killing of residual cancer cells. In recent years, due to the unique advantages of immune checkpoint inhibitors(ICIs), immunotherapy has gradually become a vital part of neoadjuvant therapy, and the scope of immunotherapy in malignant tumors expands. With administration of ICIs, revived tumor-specific CD8+ T cells proliferate and kill existing tumor cells and recirculate into the blood. After resection or ablation of the primary tumor, the remaining circulating tumor-specific CD8+ T cells and T cell clones present in the metastatic site can retain long-term anti-tumor immunity and play a vital role in continuous killing of residual cancer cells and immune surveillance. At present, the combination of targeted therapy and immune checkpoint inhibitors has achieved a higher objective response rate (ORR) and disease control rate (DCR) in the treatment of in treatment of HCC, which provides a reliable theoretical and practical basis for using as a strategy of neoadjuvant therapy.

The current reports on neoadjuvant therapy for HCC are limited to patients who are going undergo surgical resection, and there is no report on the neoadjuvant therapy prior to RFA. Since molecular targeted drugs generally have anti-angiogenic effects, drug withdrawal for two weeks or more (bevacizumab should be stopped for at least 4 weeks) before surgery is required to reduce the risk of intraoperative bleeding caused by targeted drugs and the hard-to-heal incision after operation. The longer-term drug withdrawal will prolong the preoperative waiting period, and the tumor may progress, leaving the patients loss of the opportunity for surgery. However, due to its advantage of minimal invasiveness, patients can undergo RFA directly without drug withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Research subjects understand the research content and significance, and provide the written informed consent;
* age 18 - 75 years and gender is not limited;
* a history of liver resection or RFA for HCC which was clinically or pathologically diagnosed according to the standard of the American Association for the Study of Liver Diseases; the number of lesions ≤ 3, the largest lesion ≤ 3 cm, as demonstrated on by contrast enhanced CT/MRI;
* Patients who are unable or unwilling to undergo liver resection, and have not received other anti-tumor therapies before detection of the recurrence;
* Child Pugh A (≤ 7 points), no pleural ascites and hepatic encephalopathy requiring treatment; Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-1;
* Within 7 days before enrollment, have sufficient liver and kidney function, suitable laboratory indicators (untreated): hemoglobin (HGB) ≥ 9.0 g/dl, neutrophils ≥ 1,500/mm3, PLT ≥ 50×109/L, serum ALB ≥ 28 g/L, TBIL < 50 umol/L, ALT, AST < 5 times the upper limit of normal, Bun, Cr < 1.5 times the upper limit of normal, INR < 1.7 or prolonged PT < 4 s;
* Consent to take the immune checkpoint inhibitor and molecular-targeted drugs;
* No other diseases affecting RFA treatment and targeted therapy combining with immune checkpoint inhibitors.

Exclusion Criteria:

* Patients who have a history of immune checkpoint inhibitor or targeted therapy;
* Tumor invades the branch or trunk of portal vein;
* Patients with extrahepatic metastasis;
* Patients who have an active autoimmune disease or a history of autoimmune disease, hyperthyroidism or hypothyroidism, asthma requiring bronchodilator treatment.
* Patients who have significant cardiovascular disease (heart failure grade Ⅲ or higher as defined by the New York Heart Association), myocardial infarction, unstable arrhythmia, unstable angina pectoris that occurred within 3 months before treatment;
* Patients who have a history of idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia, or an evidence of active pneumonia during chest CT scan screening;
* Patients who have received allogeneic stem cell or solid organ transplantation (including liver transplantation);
* Patients who have taken any anti-tumor Chinese herbal medicine within 7 days before enrollment;
* Patients who have any other diseases, metabolic disorders, abnormal results of physical examination or laboratory tests, which may lead to contraindication to the use of the experimental drugs, or affect the reliability of the research results, or leave the patient at high risk of treatment complications, or affect patient compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence-free survival | 1 year after treatment
  Evaluated by hepatic imaging examination (contrast-enhanced US/CT/MRI) at early stage combined with AFP and PIVKA-Ⅱtests.
1-year overall survival | 1 year after treatment
  Evaluated by hepatic imaging examination (contrast-enhanced US/CT/MRI) at early stage combined with AFP and PIVKA-Ⅱtests.

SECONDARY OUTCOMES:
procedure related complications | up to 1 year.
  procedure related complications
immune-related adverse events | up to 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of hepatobiliary surgery,Southwest Hospital, Chongqing, Chongqing Municipality, China